CLINICAL TRIAL: NCT04444154
Title: Comparison of the Effectiveness of 3 Teaching Methods in Oral Hygiene in Adolescent Orthodontic Patients: Prospective Randomized Controlled Clinical Study
Brief Title: Comparison of the Effectiveness of Three Teaching Methods in Oral Hygiene in Adolescent Orthodontic Patients
Acronym: MAHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 35RC20_8945_MAHO
Record Dates: First submitted 2020-05-12; First posted 2020-06-23 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Orthodontic Appliance
Keywords: orthodontic appliance; oral hygiene; modified orthodontic plaque index; Loë and Silness
MeSH Terms: interventions — Control Groups; Population Groups; Videotape Recording

STUDY DESIGN:
Intervention Model Description: prospective, monocentric, controlled, randomized study
Who Masked: Outcomes Assessor
Masking Description: The plaque index readings, i.e. the taking of 3 macrophotographic shots (with reflex camera, allowing the MOP plaque index to be assessed in a second step), and the clinical index of gingival inflammation will be performed at each appointment (except during the dedicated session of group 3) by an examiner who will be blind from the group belonging to each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): oral hygiene advice given orally
  Interventions: Behavioral: Control group
- Group with active participation (Active Comparator): oral hygiene advice given orally and demonstration of brushing methods in the sink with active participation
  Interventions: Behavioral: Group with active participation
- Group with video and quizz (Experimental): oral hygiene advice given orally and an additional appointment between the device bonding appointment and the first check-up. This is a 15-minute session dedicated to teaching oral hygiene. This session will include watching of an educational video followed by a quiz, as well as the application of the methods taught in the sink (using plate developer and the Oral B electric toothbrush with special orthodontic head).
  Interventions: Behavioral: Group with video and quizz

INTERVENTIONS:
Behavioral: Control group — oral hygiene advice given orally in the chair during the bonding appointment and at each check-up appointment.
  Arms: Control group
Behavioral: Group with active participation — oral hygiene advice given orally in the chair during the bonding appointment and at each check-up appointment with a demonstration of brushing methods in the sink with active participation (use of plate developer and then the Oral B electric toothbrush with special orthodontic head) during the bonding appointment as well than at each check-up appointment.
  Arms: Group with active participation
Behavioral: Group with video and quizz — oral hygiene advice given orally in the chair during the bonding appointment and at each check-up appointment with have an additional appointment between the device bonding appointment and the first check-up. This is a 15-minute session dedicated to teaching oral hygiene. This session will include watching of an educational video followed by a quiz, as well as the application of the methods taught in the sink (using plate developer and the Oral B electric toothbrush with special orthodontic head).
  Arms: Group with video and quizz

SUMMARY:
Orthodontic appliances have been shown to interfere with oral hygiene maneuvers by providing many additional sites for formation and retention of biofilm.

Its accumulation is responsible for undesirable effects such as decays and periodontal pathologies. These lower the benefit / risk ratio of orthodontic treatments. In addition, their management is not negligible at the macroeconomic level.

As such, it is more than necessary for the orthodontist to teach oral hygiene methods adapted to each of his patients fitted to limit the risk of appearance of biofilm.

DETAILED DESCRIPTION:
Patients applying for orthodontic treatment with braces in the orthodontic unit of the Rennes dental center will be offered to participate in the study. For each patient, the inclusion and non-inclusion criteria will be checked, and consent and a document explaining the course of the study will be delivered to them personally. The duration of the study will be 6 months for each of them. Each will be randomized to one of three study groups. Throughout the study, patients in groups 1 and 2 will have to make 5 appointments. Group 3 patients must honor 6 appointments.

Patients in group 1 (control group) will receive oral hygiene advice given orally in the chair during the bonding appointment and at each check-up appointment. Patients in group 2 will receive these same oral advice, associated with a demonstration of brushing methods in the sink with active participation (use of plate developer and then the Oral B electric toothbrush with special orthodontic head) during the bonding appointment as well than at each check-up appointment. Patients in group 3 will receive the same treatment as those in group 1 but will have an additional appointment between the device bonding appointment and the first check-up. This is a 15-minute session dedicated to teaching oral hygiene. This session will include watching of an educational video followed by a quiz, as well as the application of the methods taught in the sink (using plate developer and the Oral B electric toothbrush with special orthodontic head).

At the end of the appliance bonding appointment (first appointment) each patient (from each group) will leave with a hygiene kit including an electric toothbrush with two orthodontic heads, an Oral B toothpaste, from orthodontic wax and the analgesic prescription conventionally performed when installing a device.

The plaque index readings, i.e. the taking of 3 macrophotographic shots (with reflex camera, allowing the MOP plaque index to be assessed in a second step), and the clinical index of gingival inflammation will be performed at each appointment (except during the dedicated session of group 3) by an examiner who will be blind from the group belonging to each patient.

Exception made for the day of bonding, during which the plate index reading will be made just before the placement of the multi fasteners via the Loë and Silness plate index (which is an index adapted to patients not fitted).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 11 to 17 * years;
* Patient with stable adolescent teeth, young adult or adult teeth;
* Requiring a fixed orthodontic treatment without extraction (other than wisdom teeth) at least to the maxillary arch;
* Affiliated, himself or through his parents to a social security scheme;
* Having received information on the protocol and having given free, informed and written consent.
* Whose holders of parental authority have received information on the protocol and have given free, informed and written consent.

  * Aged under 18 at the end of the 6 months of participation

Exclusion Criteria:

* Patient with periodontal disease or progressive carious lesions;
* Patient with a prosthetic crown or composite restoration on the central and / or lateral maxillary incisor;
* Patient with systemic disease, major syndrome or cleft palate;
* Patient with an abnormal dental structure (eg fluorosis, MIH, imperfect amelogenesis, etc.);
* Patients taking long-term medication influencing periodontal health (corticosteroids, anti-epileptics, etc.);
* Patient with a physical or mental handicap preventing him from carrying out oral hygiene maneuvers independently;
* Patient refusing to use the products and instruments prescribed for the study;
* Patients with dental agenesis;
* Patients with poor command of the French language
* Patient deprived of liberty by judicial or administrative decision or subject to a legal protection measure;
* Pregnant patient;
* Smoking patient.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-01-29 (Actual); Primary Completion 2025-01-29 (Estimated); Study Completion 2025-01-29 (Estimated)

PRIMARY OUTCOMES:
Compare the effectiveness of 3 methods of teaching oral hygiene in terms of controlling biofilm formation: MOP (Modified Orthodnotic Plaque Index) classification | 6 months of intervention
  The average plaque index at six months after inclusion according to the MOP (Modified Orthodnotic Plaque Index) classification. It is evaluated on macro photography in a standardized manner by a blind examiner of the patient's randomization arm. The values range from 0 to 4 for each tooth, which makes an average score of 0 to 48 for the maxillary arch. 0 is the absence of plaque while 48 is an abundance of plaque on all teeth, the worst situation. The score is expressed in absolute value without unit.

SECONDARY OUTCOMES:
Compare the effectiveness of three teaching methods in oral hygiene for the control of gum inflammation: gingival index at six months after inclusion according to the Loë and Silness scale | 6 months after bonding the device.
  The mean gingival index at six months after inclusion according to the Loë and Silness scale. It will be evaluated in the mouth in a standardized manner by a blind examiner of the patient's randomization arm. The values range from 0 to 3 for each side of each tooth, which makes an average score of 0 to 144 for the maxillary arch. 0 corresponds to no bleeding on probing whereas 3 characterizes a situation of spontaneous bleeding of the gum, worst situation. The score is expressed in absolute value without unit.
Compare the effectiveness of three methods of teaching oral hygiene over time: MOP classification plate index | J0 (during the installation of the device)
  The comparison of the three treatment groups as a function of time will be based on two judgment criteria. The first is the MOP classification plate index. It is evaluated on macrophotographs in a standardized manner by a blind examiner of the patient's randomization arm. The values range from 0 to 4 for each tooth, which makes an average score of 0 to 48 for the maxillary arch. 0 is the absence of plaque while 48 is an abundance of plaque on all teeth, the worst situation. The score is expressed in absolute value without unit.
Compare the effectiveness of three methods of teaching oral hygiene over time: gingival index according to the Loë and Silness scale | J0 (during the installation of the device)
  The comparison of the three treatment groups as a function of time will be based on two judgment criteria. The second is the gingival index according to the Loë and Silness scale. It will be evaluated in the mouth in a standardized manner by a blind examiner of the patient's randomization arm. The values range from 0 to 3 for each side of each tooth, which makes an average score of 0 to 144 for the maxillary arch. 0 corresponds to no bleeding on probing whereas 3 characterizes a situation of spontaneous bleeding of the gum, worst situation. The score is expressed in absolute value without unit.
Compare the effectiveness of three methods of teaching oral hygiene over time: MOP classification plate index | at 1½ months after installation of the device
  The comparison of the three treatment groups as a function of time will be based on two judgment criteria. The first is the MOP classification plate index. It is evaluated on macrophotographs in a standardized manner by a blind examiner of the patient's randomization arm. The values range from 0 to 4 for each tooth, which makes an average score of 0 to 48 for the maxillary arch. 0 is the absence of plaque while 48 is an abundance of plaque on all teeth, the worst situation. The score is expressed in absolute value without unit.
Compare the effectiveness of three methods of teaching oral hygiene over time: gingival index according to the Loë and Silness scale | at 1½ months after installation of the device
  The comparison of the three treatment groups as a function of time will be based on two judgment criteria. The second is the gingival index according to the Loë and Silness scale. It will be evaluated in the mouth in a standardized manner by a blind examiner of the patient's randomization arm. The values range from 0 to 3 for each side of each tooth, which makes an average score of 0 to 144 for the maxillary arch. 0 corresponds to no bleeding on probing whereas 3 characterizes a situation of spontaneous bleeding of the gum, worst situation. The score is expressed in absolute value without unit.
Compare the effectiveness of three methods of teaching oral hygiene over time: MOP classification plate index | at 3 months after installation of the device
  The comparison of the three treatment groups as a function of time will be based on two judgment criteria. The first is the MOP classification plate index. It is evaluated on macrophotographs in a standardized manner by a blind examiner of the patient's randomization arm. The values range from 0 to 4 for each tooth, which makes an average score of 0 to 48 for the maxillary arch. 0 is the absence of plaque while 48 is an abundance of plaque on all teeth, the worst situation. The score is expressed in absolute value without unit.
Compare the effectiveness of three methods of teaching oral hygiene over time: gingival index according to the Loë and Silness scale | at 3 months after installation of the device
  The comparison of the three treatment groups as a function of time will be based on two judgment criteria. The second is the gingival index according to the Loë and Silness scale. It will be evaluated in the mouth in a standardized manner by a blind examiner of the patient's randomization arm. The values range from 0 to 3 for each side of each tooth, which makes an average score of 0 to 144 for the maxillary arch. 0 corresponds to no bleeding on probing whereas 3 characterizes a situation of spontaneous bleeding of the gum, worst situation. The score is expressed in absolute value without unit.
Compare the effectiveness of three methods of teaching oral hygiene over time: MOP classification plate index | at 4½ months after installation of the device
  The comparison of the three treatment groups as a function of time will be based on two judgment criteria. The first is the MOP classification plate index. It is evaluated on macrophotographs in a standardized manner by a blind examiner of the patient's randomization arm. The values range from 0 to 4 for each tooth, which makes an average score of 0 to 48 for the maxillary arch. 0 is the absence of plaque while 48 is an abundance of plaque on all teeth, the worst situation. The score is expressed in absolute value without unit.
Compare the effectiveness of three methods of teaching oral hygiene over time: gingival index according to the Loë and Silness scale | at 4½ months after installation of the device
  The comparison of the three treatment groups as a function of time will be based on two judgment criteria. The second is the gingival index according to the Loë and Silness scale. It will be evaluated in the mouth in a standardized manner by a blind examiner of the patient's randomization arm. The values range from 0 to 3 for each side of each tooth, which makes an average score of 0 to 144 for the maxillary arch. 0 corresponds to no bleeding on probing whereas 3 characterizes a situation of spontaneous bleeding of the gum, worst situation. The score is expressed in absolute value without unit.

CONTACTS AND LOCATIONS:
Overall Officials: Damien BREZULIER, Dr, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU de RENNES, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Fouler A, Jeanne S, Sorel O, Brezulier D. How effective are three methods of teaching oral hygiene for adolescents undergoing orthodontic treatment? The MAHO protocol: an RCT comparing visual, auditory and kinesthetic methods. Trials. 2021 Feb 15;22(1):144. doi: 10.1186/s13063-021-05093-z. PMID 33588930